CLINICAL TRIAL: NCT06732388
Title: Repurposing Itraconazole for Secondary Prevention of Metaplasia and Primary Prevention of Cancer in Patients With High-Risk Barrett's Esophagus in Combination With Ablation
Brief Title: Itraconazole in Combination With Ablation for the Prevention of Esophageal Cancer in Patients With High-risk Barrett's Esophagus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCI-2024-10070; NCI-2024-10070 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UMI23-16-01 (Other: University of Michigan Rogel Cancer Center); UMI23-16-01 (Other: DCP); P30CA046592 (NIH); UG1CA242632 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2024-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Barrett Esophagus; Clinical Stage I Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIA Esophageal Adenocarcinoma AJCC v8; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Biopsy; Specimen Handling; Endoscopy; Itraconazole; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants as well as the study team will be blinded to the study drug assignment. The study endoscopist will be blinded to the treatment group to avoid bias. Will ensure that the laboratory personnel running the assays are blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (itraconazole) (Experimental): Patients receive itraconazole PO twice daily (BID) on days 1-42 of each cycle. Cycles repeat every 6 weeks for up to 2 cycles as long as there is an absence of disease progression or unacceptable toxicity. Patients undergo usual standard of care endoscopy and radiofrequency ablation on study. Patients also undergo blood sample collection throughout the study as well as tissue biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Endoscopic Procedure; Drug: Itraconazole; Other: Questionnaire Administration; Procedure: Radiofrequency Ablation
- Group II (placebo) (Placebo Comparator): Patients receive placebo PO BID on days 1-42 of each cycle. Cycles repeat every 6 weeks for up to 2 cycles as long as there is an absence of disease progression or unacceptable toxicity. Patients undergo usual standard of care endoscopy and radiofrequency ablation on study. Patients also undergo blood sample collection throughout the study as well as tissue biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Endoscopic Procedure; Drug: Placebo Administration; Other: Questionnaire Administration; Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Endoscopic Procedure — Undergo endoscopy
  Other Names: Endoscopic Examination; Endoscopy; ES
Drug: Itraconazole — Given PO
  Other Names: Lozanoc; Oriconazole; R 51,211; Sporanox
  Arms: Group I (itraconazole)
Drug: Placebo Administration — Given PO
  Arms: Group II (placebo)
Other: Questionnaire Administration — Ancillary studies
Procedure: Radiofrequency Ablation — Undergo radiofrequency ablation
  Other Names: Ablation, Radiofrequency; Radiofrequency Interstitial Ablation; RFA

SUMMARY:
This phase II trial tests how well itraconazole works in combination with the usual standard of care endoscopy with ablation for the prevention of esophageal cancer in patients who have high-risk Barrett's esophagus (BE). BE is a condition in which the lining of the esophagus changes and becomes more like the tissue that lines the intestine. People with Barrett's esophagus have a higher risk of developing esophageal cancer. Itraconazole is a drug used to prevent or treat fungal infections. Ablation refers to the removal of abnormal tissue using heat. Endoscopy is a procedure for looking at the esophagus using a long, flexible tube called an endoscope, which has a video camera at the end. Radiofrequency ablation is a type of heat therapy that uses radiofrequency energy (similar to microwave heat) to destroy the abnormal tissue in the esophagus. Giving itraconazole in combination with standard of care endoscopy with ablation may improve the effects of ablation and prevent esophageal cancer in patients with high-risk Barrett's esophagus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate if itraconazole in the peri-ablation period in participants with high-risk Barrett's esophagus (BE) can accelerate BE regression i.e., achieve complete resolution of intestinal metaplasia (CRIM) faster than the control group.

SECONDARY OBJECTIVES:

I. To measure the time to event of complete eradication of dysplasia (CED). II. To measure the rate of BE recurrence during routine follow-up. III. To determine the safety and tolerability of itraconazole in participants with high-risk BE.

IV. To correlate levels of itraconazole and its primary metabolite hydroxyitraconazole in plasma and esophageal tissues with treatment response.

V. To compare biosocial impact on the participants in the itraconazole and control arms.

EXPLANATORY OBJECTIVE:

I. To correlate the degree of inhibition of Hedgehog (Hh), PI3K-AKT, and VEGFR2 signaling pathways with treatment response.

EXPLORATORY OBJECTIVES:

I. To determine whether expression (baseline and magnitude of change) of stem cell markers such as LGR5/CD44/DCAMKL1 can predict treatment response.

II. To bank blood samples and tissue biopsies for future analyses to understand the determinants of response.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive itraconazole orally (PO) twice daily (BID) on days 1-42 of each cycle. Cycles repeat every 6 weeks for up to 2 cycles as long as there is an absence of disease progression or unacceptable toxicity. Patients undergo usual standard of care endoscopy and radiofrequency ablation on study. Patients also undergo blood sample collection throughout the study as well as tissue biopsy on study.

GROUP II: Patients receive placebo PO BID on days 1-42 of each cycle. Cycles repeat every 6 weeks for up to 2 cycles as long as there is an absence of disease progression or unacceptable toxicity. Patients undergo usual standard of care endoscopy and radiofrequency ablation on study. Patients also undergo blood sample collection throughout the study as well as tissue biopsy on study.

After completion of study treatment, patients are followed up at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with history of prior esophagogastroduodenoscopy (EGD) with an established diagnosis of BE ≥ 2 cm with either low-grade dysplasia (LGD) or high-grade dysplasia (HGD) or T1a esophageal adenocarcinoma (EAC), naïve to treatment, and being considered for ablation.

  * Note: An eligible diagnosis from an EGD outside of the enrollment sites is allowed for inclusion as long as the biopsies have been reviewed by two pathologists. The two pathologists could include a pathologist from the referring site and an institutional pathologist at the local enrolling site, two pathologists from the referring site, or two pathologists from the local enrolling site. The diagnosis between two pathologists has to be concordant regarding the presence of dysplasia or cancer. Discrepant diagnoses will be resolved by a third pathologist, if needed
* Participants older than 18 years will be enrolled. Because the incidence of BE and related cancer is very low in participants < 18 years of age, children are excluded from this study
* Clinically eligible for EGD and endoscopic treatment of BE
* Absolute neutrophil count ≥ 1,000/microliter
* Platelets ≥ 100,000/microliter
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)

  * Note: Higher total bilirubin levels (≤ 3 mg/dL) can be allowed if due to known benign liver condition, i.e. Gilbert's
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) ≤ 1.5 × institutional upper limit of normal
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Participants on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible
* There are no controlled data on the effects of itraconazole on the developing human fetus at the recommended therapeutic dose. For this reason and because azoles are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) two months prior to study entry, for the duration of study participation and two months after completing the study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current New York Heart Association (NYHA) class III or IV congestive heart failure
* Prolonged corrected QT (QTc) (> 450 ms for men and > 470 ms for women)
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to itraconazole
* Uncontrolled intercurrent illness., or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because itraconazole is a class C agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with itraconazole, breastfeeding should be discontinued if the mother is treated with itraconazole
* Critical drug interactions (grades D or higher) with other medications metabolized by cytochrome P450(CYP)3A4 (if the medication cannot be discontinued or switched or dose modified); these decisions will be made on a case-by-case basis by the site investigators in consultation with the treating provider. Drug interactions can be assessed using one of the available on-line resources, for instance, UpToDate or Clinical Formulary and/or in collaboration with a clinical pharmacist.

  * Note: If there are potential drug interactions that do not exclude the participant from the study, a brief research note summarizing the decision-making process about potential drug interactions and their management will be required before the participants are enrolled in the trial
* History of eosinophilic esophagitis
* History of strictures not allowing passage of the radiofrequency ablation (RFA) assembly
* Participants must not have evidence of active/recurrent invasive cancer of a non-esophageal organ
* Participants with EAC greater than stage T1a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Time to complete resolution of intestinal metaplasia (CRIM) in days | Between day 1, cycle 1 (1 cycle = 6 weeks) and the date of endoscopy at which the participant is deemed to reach CRIM
  CRIM will be defined based on the absence of visible Barrett's esophagus (BE) and invisible BE (i.e., no intestinal metaplasia [IM] in biopsies of the gastroesophageal junction and the cardia). Will be reported descriptively. Will compare the unadjusted hazard rates between the itraconazole and control groups using log rank test.

SECONDARY OUTCOMES:
Time to complete eradication of dysplasia | Between day 1, cycle 1 (1 cycle = 6 weeks) and the date of endoscopy at which surveillance biopsies do not show dysplasia
  Will be assessed by surveillance biopsies at the time of the endoscopy that documents CRIM and the biopsies at the time of first surveillance endoscopy will be evaluated for dysplasia.
Rate of BE recurrence over follow-up | At 12 months after CRIM
  Will be assessed between the study treatment group and the control group. BE recurrence will be defined as histologic presence of IM (with or without dysplasia) in biopsies from the tubular esophagus or in biopsies at the gastroesophageal junction. The results from the standrd of care endoscopy closest to the 12-month time point after CRIM will be used to collect information for this endpoint.
Incidence of adverse events | Up to 30 days after the end of intervention
  Will be assessed by National Cancer Institutes Common Terminology Criteria for Adverse Events version 5.0 criteria to document adverse events and measure specific laboratory parameters to monitor for the safety and tolerability of itraconazole and assessed by descriptive statistics.
Correlate levels of itraconazole and its primary metabolite hydroxyitraconazole | After two weeks of itraconazole
  Will be assessed in plasma and esophageal tissues with treatment response. Will measure these metabolites after two weeks of itraconazole therapy by obtaining biopsies of the esophagus. These measurements will be correlated with biomarker and clinical response to understand how tissue levels of the drug change the molecular and primary endpoints. Will also measure the blood levels to test the feasibility of blood levels for prediction of clinical response in the future.
Biosocial impact | At baseline and at the end of the study
  Will be assessed by questionnaires to collect information about the biosocial endpoints. These will include cancer-specific distress questionnaire, Gastrointestinal Symptom Rating Scale, Health-Related Quality of life short form 12 version 2, and Patient-Reported Outcomes Measurement Information System anxiety and depression scores as previously used at the beginning and at the end of the study. The summary measures such as mean or median of these distress scores will be compared between arms using t-test (or Wilcoxon rank test in case of non normality). Linear regression models will be used for studying the differences in the average distress scores between arms adjusted for age, sex and prior history of anxiety or depression.

OTHER OUTCOMES:
Correlation of the degree of inhibition of Hh, PI3K-AKT, and VEGFR2 signaling pathways with treatment response | After two weeks of study drug administration
  Measures will be assessed in biopsies of the gastroesophageal junction as well as in biopsy of BE after two weeks of study drug administration by histological techniques.
Expression of cancer stem cell markers such as LGR5/CD44/DCAMKL1 | After two weeks of itraconazole
  Measures will be assessed in biopsies of the gastroesophageal junction as well as biopsies of BE after two weeks of study drug administration by histological techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Bansal, MD, Principal Investigator — University of Kansas Medical Center
Locations (6):
- United States (6):
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm